CLINICAL TRIAL: NCT01488006
Title: 5- Year Follow-up in Total Shoulder Arthroplasty for Primary Glenohumeral Osteoarthritis: A Prospective Multicenter Study
Brief Title: Columbia Shoulder Study (CSS)
Acronym: CSS
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: AAAA5360
Record Dates: First submitted 2011-11-29; First posted 2011-12-08 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Osteoarthritis of Glenohumeral Joint
Keywords: Primary Glenohumeral Osteoarthritis; Total shoulder arthroplasty; Total shoulder replacement; Osteoarthritis; Multicenter study
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bigliani/Flatow Shoulder System: Other than the Bigliani/Flatow device, there will be no difference in treatment between those patients undergoing arthroplasty with the Bigliani / Flatow prosthesis and those who previously received other prosthesis. APatients who decide to participate in the study will complete various forms prior to surgery (The Informed Consent, Contact Information Form, Demographics Module, and standard outcomes forms such as American Shoulder and Elbow Surgeon Score form, Constant's Score form, and the Simple Shoulder Test, EuroQOL and SF-36). The patient will also complete forms postoperatively at 3-month, 6-month, 1-year, 2-year, 3-year, 4-year and 5-year intervals (American Shoulder and Elbow Surgeon Score form, Constant's Score form, Simple Shoulder Test, EuroQOL and SF-36).
  Interventions: Device: Bigliani/Flatow Shoulder System

INTERVENTIONS:
Device: Bigliani/Flatow Shoulder System — Primary Total Shoulder Arthroplasty with the Bigliani/Flatow prosthesis

SUMMARY:
This prospective study will evaluate the Bigliani/Flatow prosthesis. The aims of this study are to establish the safety, effectiveness, and value of the prosthetic system, and to collect information from expert shoulder surgeons as to features of the implants, instruments, and techniques which may be further improved. In this study, the investigators hypothesize that this prosthetic device will significantly improve long-term patient-based outcomes, functional status and quality of life.

DETAILED DESCRIPTION:
Over the last two decades, total shoulder joint replacement - or arthroplasty - has become a commonly performed procedure for the treatment of painful arthritis of the shoulder, and numerous studies have demonstrated its success. During this time, much has been learned about the efficacy, as well as the complications, of the procedure, and since its introduction in the 1950's, shoulder arthroplasty has undergone an evolution in design. The value of such innovations has not yet been determined and will depend on the results of long term follow-up studies. The purpose of this study is to provide follow-up information and design modification directives.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or over.
* Patient must have signed The Informed Consent and Release of Medical Information forms.
* The patient can be a man, postmenopausal woman, or a woman who is likely to become pregnant but is using adequate contraceptive precautions (defined as oral contraceptives, intrauterine devices, surgical contraception or a combination of a condom and spermicide).
* Patient needs a total shoulder arthroplasty (humeral head and glenoid).
* Patient has a diagnosis of primary osteoarthritis.

Exclusion Criteria:

* Obstacles, which pose an inordinately high surgical risk, in the judgment of the certified surgeon.
* Class IV or higher anesthetic risk.
* Patient has a recent history of psychiatric disease (including drug or alcohol abuse) that is likely to impair the compliance with the study protocol.
* Patient has had a shoulder fracture.
* Patient had previous shoulder surgeries with the exception of an arthroscopic debridement procedure.
* The patients has a massive rotator cuff tear (rupture >3 cm or total cicatrisation) demonstrated at time of the surgery that precludes the total shoulder replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited when the decision to undergo shoulder arthroplasty is made. The surgeon will confirm that the subject is appropriate for inclusion in the study. The surgeon will confirm that the subject is appropriate for inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2001-04; Primary Completion 2009-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Preoperative Radiographic Measurements of Standard Glenohumeral Relationships | Up to 16 weeks prior to date of surgery
Change in Post-operative Radiographic Measurements of Prosthetic Relationships (Anteroposterior and Axillary x-rays) | Up to 5 years postoperatively
  Measurements include acromiohumeral interval, head to tuberosity distance, coracoid to glenohumeral joint distance, coracoid to tuberosity distance, humeral stem position (valgus/varus), humeral congruity and subluxation, glenoid comp version.
Change in Radiographic Analysis for Lucent Lines and Prosthesis Loosening | Up to 5 year postoperatively
  glenoid and humeral component lucency

SECONDARY OUTCOMES:
Change in Score on Short-Form 36 (SF-36) | Up to 5 years postoperatively.
  Mental component score, physical component score, mental health, physical function, role emotional, role physical, social function, vitality, bodily pain and general health
Change in Score on EuroQOL (EQ-5D) | Up to 5 years postoperatively.
  Total index, visual analog scale, mobility, anxiety/depression, pain/discomfort, self-care, and usual activities.
Change in ASES (American Shoulder and Elbow Surgeons) Score | Up to 5 years postoperatively.
Change in Total Score on Simple Shoulder Test (SST) | Up to 5 years postoperatively.
  Total score.
Change in Constant Score | Up to 5 years postoperatively.
Change in Range of Motion | Up to 5 years postoperatively.
  Active and passive external rotation at 90 degrees and at side, active and passive forward elevation, active and passive abduction, active and passive internal rotation

CONTACTS AND LOCATIONS:
Overall Officials: William N Levine, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States